CLINICAL TRIAL: NCT06615908
Title: A Randomized Double-blinded Controlled Trial for the Treatment of Persisting Symptoms After Concussion With Psilocybin-assisted Therapy: A Safety and Feasibility Trial
Brief Title: Treatment of Persisting Symptoms After Concussion With Psilocybin Assisted Therapy
Acronym: PatACT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB24-0334
Record Dates: First submitted 2024-09-11; First posted 2024-09-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-05

CONDITIONS: Persisting Symptoms After Concussion
Keywords: Psychotherapy; Psilocybin; Concussion; Mild Traumatic Brain Injury; Acceptance and Commitment Therapy
MeSH Terms: conditions — Brain Concussion | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The group assignments to active (25mg) and control (1mg) psilocybin-assisted therapy will be based on a blocked randomization list (10 participants per block) using sealed envelopes created by an employee of the University of Calgary, who will not be involved in the conduct, or the analysis of the study.
  The pharmacy administering the psilocybin will be responsible for maintaining the master randomization code list and only the technician preparing the samples will have access to the envelopes and code list.
  When a new study ID is generated, the technician is to verify the randomization and prepare the participant's study intervention accordingly. Unblinding will only occur once the entire study is completed, and the database has been locked.
  The trials active intervention and comparator will be provided by the manufactures and will be identical in shape, colour, and weight.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose (25mg) (Experimental): High Dose (25mg) PEX010 (Oral Psilocybin), 25mg; single dose (20 participants) administered 24hrs prior to first ACT session
  Interventions: Drug: Psilocybin
- Low dose (1mg) (Active Comparator): Low Dose (1mg) PEX010 (Oral Psilocybin), 1mg; single dose (20 participants)administered 24hrs prior to first ACT session
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — See treatment arm description.
  Other Names: magic mushrooms; PEX010

SUMMARY:
The goal of this randomized controlled trial is to evaluate the safety, feasibility, and efficacy of psilocybin assisted therapy as an intervention to reduce symptom burden in adult patients (aged 18-65) with persisting symptoms after concussion (PSaC).

This trail will test the following 2 aims:

AIM 1 : To test the safety and feasibility of an active psilocybin-assisted psychotherapy to an active control for patients with PSaC.

AIM 2: To evaluate the efficacy of an active psilocybin-assisted psychotherapy compared to an active control as a treatment for PSaC.

Participants will be asked to:

* Complete a 2-part screening process
* Attend a baseline assessment
* Complete a psychoeducation preparation session(s)
* Attend psilocybin administration session (receive high dose [25mg] or low dose psilocybin [1mg])
* Complete 5 weekly sessions of Acceptance and commitment therapy (ACT)
* Repeat outcome measures at 1-week, 4 weeks, 3 months, and 6 months post-psilocybin administration (online only at 6 months).

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the safety, feasibility, and efficacy of psilocybin assisted therapy administered with Acceptance and Commitment Therapy (ACT) as an intervention to reduce symptom burden in patients with persisting symptoms after concussion (PSaC).

This trail will test the following 2 aims:

AIM 1 : To test the safety and feasibility of an active/high dose (25mg) psilocybin-assisted psychotherapy to an active control (1mg) for adults with PSaC. Safety will be determined through the reporting of adverse events and response following psilocybin for each participant up to 6-months. Feasibility will be determined through recruitment, enrollment, and adherence rates.

AIM 2: To evaluate the efficacy of an active/high dose (25mg) psilocybin-assisted psychotherapy compared to an active control (1mg) as a treatment for PPCS at 1-week, 4 weeks, 3 months, and 6 months post-psilocybin administration. The primary efficacy outcome will be the change in PSaC burden (RPQ).

The secondary efficacy outcomes will include measures of headache, dizziness, mood, anxiety, post-traumatic stress, cognitive flexibility, emotional regulation, and quality of life.

A total of 40 male and female patients between the ages of 18-65 with a diagnosis of mild traumatic brain injury (American College of Rehabilitation Medicine 2023 criteria) who meet criteria for persisting symptoms after concussion (ICD-10) within 3 months to 5 years will be recruited from Calgary brain injury clinics and the community.

All patients will undergo a thorough, 2-part screening procedure. Eligible participants will be randomly allocated 1:1 to either the high dose (20 participants) or low dose (20 participants) psilocybin groups. All participants will be asked to attend a baseline session consisting of clinical and behavioural outcome measures, followed by a pre-dosing psychoeducation session. Following the single dosing session, participants will complete 5 weekly ACT sessions. Outcome measure assessments will be repeated at 1-week, 4 weeks, 3 months, and 6 months post-dosing.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Individuals of all sexes, gender identities, and ethnicities
* Ages 18 to 65 years at the time of screening
* Diagnosis of concussion based on the 2024 ACRM criteria
* Meet ICD-10 criteria for PSaC for at least 3-months to a maximum of 5 years
* Have an overall RPQ score ≥ 13 with 3 or more symptoms scored ≥3
* Limited lifetime use of serotonergic hallucinogens
* Ability to read/write English

An individual who meets any of the following criteria will be excluded from participation in this study:

* Severe or moderate substance use disorder other than nicotine in past 6 months
* Lifetime diagnosis of schizophrenia or bipolar disorders (or first or second-degree relative)
* Active suicidal ideation or serious attempt within the past 1 year.
* Current pregnancy or nursing, trying to become pregnant
* Any notable abnormality on ECG or routine medical blood laboratory test
* Insulin-dependent diabetes; if taking oral hypoglycemic agent, then no history of hypoglycemia
* Epilepsy with a history of seizures
* Current or recent (within 12 weeks) participation in a clinical trial
* Cognitive impairment (SLUMS score <20)
* Suffered a moderate/severe TBI at least once in lifetime
* Any other circumstances that, in the opinion of the investigators, compromises participant safety

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Throughout study completion, an average of 6 months
  Safety will be determined based on adverse reactions and symptom reporting (categorized as mild, moderate, and severe)
Study protocol efficacy | Throughout study completion, an average of 6 months
  The primary efficacy outcome is the Rivermead Post-Concussion Symptoms Questionnaire (RPQ).The RPQ assesses the severity of 16 commonly experienced PSaC symptoms using a scale of 0 ("not experienced") to 4 ("severe problem"), with higher scores indicating greater PSaC symptom burden.
Study protocol feasibility | Screening, enrolment, intervention, and participation up to study end point (6-months)
  The feasibility will be determined based on recruitment (greater than 30% of those screened eligible), attendance (70% intervention appointment attendance), retention (70% complete study protocol)

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale Self report (MADRS-S) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  The MADRS is a 10-item assessment of depressive symptoms using a recall period of the past 7 days. Total scores range from 0-60, with higher scores indicating greater depression.
Generalized Anxiety Disorder-7 (GAD-7). | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  The GAD-7 is a 7-item tool which assess anxiety. Individuals rate how often they have been bothered by seven listed problems and score their responses from 0 ("not at all") to 3 ("nearly every day"). Total scores for anxiety severity are: 0-4: minimal anxiety; 5-9: mild; 10-14: moderate; 15-21: severe anxiety.
Sleep and Concussion Questionnaire (SCQ) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  During the SCQ-initial, participants use the timeframe of the 6-months prior to the concussion, and since the concussion. The SCQ-follow-up will have a recall period of since the most recent SCQ was completed. Total scores of 0-7 indicate no clinically significant change; 8-15: subclinical change; 16-22: clinical changes of moderate severity; 23-36: clinically severe changes in sleep or wakefulness.
Headache Impact Test (HIT-6). | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  This 6-item tool assesses how headache intensity impacts daily life functioning. Headache intensity and frequency are measured from "never" to "always", with greater scores indicating greater impact on daily life function due to headache. Total scores of 49 or less indicate headaches have little to no impact on daily life; 50-55: headaches have some impact on life; 56-59: headaches have substantial impact on life; 60 or more: headaches have severe impact on life.
Dizziness Handicap Questionnaire (DHI) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  A 25-item self-reported questionnaire which assesses the impact of dizziness on daily life. Scores from functional, emotional, and physical domains are summed to give a score between 0-100 with greater scores indicating greater impact.
PTSD Checklist for DSM-5 (PCL-5) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  A 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Greater symptom scores indicate greater symptom burden
The Quality of Life after Brain Injury (QOLIBRI) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  This questionnaire measures health-related quality of life specific to individuals after traumatic brain injury. Covers six domains of health-related quality of life (cognition, self, daily life and autonomy, social relationships, emotions, and physical problems) to provide an overall score, with higher scores indicating greater quality of life.
Difficulties in Emotion Regulation Scale (DERS) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  A 36-item self-report scale designed to assess multiple aspects of emotion dysregulation. Six subscale scores and a total score are calculated.
Think Aloud Task | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, and 3 months post-dosing]
  The Thinking Aloud Task (TAT) measures cognitive flexibility in relation to thought dynamics, tapping into the speed and expansiveness of thoughts, which relate to real-time emotion regulation and overall social and emotional well-being.
Probabilistic Reversal Learning Task | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, and 3 months post-dosing]
  The Probabilistic Reversal Learning (PRL) task is a measure of reward-related cognitive flexibility that requires participants to choose a shape that fits an inferred rule and adapt behavior once rules switch
The Acceptance and Action Questionnaire II (AAQ-II) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  A 7-item questionnaire measuring psychological flexibility. Scores range from 0 to 49 with higher scores indicating greater psychological flexibility
The Acceptance and Action after Brain Injury Questionnaire (AAQ-ABI) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  A 7-item questionnaire which measures psychological flexibility about the thoughts and feelings related to brain injury. Scored on a 5-point Likert scale, scores range from 0-36 with higher scores indicating greater psychological flexibility
Cognitive Fusion Questionnaire (CFQ-7) | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, 3 months, and 6 months post-dosing]
  A 7-point Likert scale measuring cognitive fusion. Scores range from 0 to 49 with higher scores indicating greater fusion with one's thoughts.
Bergs Card Sorting Task | Throughout study completion, an average of 6 months [assessed at baseline, and 1-week, 4 weeks, and 3 months post-dosing]
  Cognitive flexibility task - Participants must select the stimulus that is different from others based on feedback and adapt their responses once the criteria for correct choice switches. Perseverative errors are defined as the number of instances in which three incorrect responses are made based on a previous rule, and they are thought to reflect less cognitive flexibility (or cognitive rigidity)

CONTACTS AND LOCATIONS:
Overall Officials: Chantel T Debert, MD MSc FRCPC, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No